CLINICAL TRIAL: NCT02026674
Title: Reliability of Home Uroflowmetery Using a Disposable Digital Device in Comparison to Standard Clinical Uroflowmetry in Men With LUTS
Brief Title: Reliability of Home Uroflowmetery Using a Disposable Digital Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Flometrica Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLO-ISR-01
Record Dates: First submitted 2013-12-24; First posted 2014-01-03 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: urineflow; luts; urine flow; uroflometry; bph
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FloRite (Experimental): LUTS patients that used FloRite for home urine flow diagnostics.
  Interventions: Device: FloRite

INTERVENTIONS:
Device: FloRite — Disposable home use urine flow meter.

SUMMARY:
The FloRite™ device is a disposable urine flow meter, indicated for use in a home setting.

The device provides Urofowmetry measurements, similar to clinic's measurements. Clinic-based uroflowmetry has some flaws; the setting is artificial and often it is difficult to void at the desired moment. Moreover, a single measurement of the voided parameters is a poor representative of the patient condition due to high variability of the measured parameters. Performing multiple Urofowmetry measurements provides representative and more accurate results, in a more patient-friendly, cost effective method.

DETAILED DESCRIPTION:
The FloRite™ product is a disposable urine flow meter. The patient needs to urinate into the device and at the end of urination the patient needs to disconnect a USB drive from the device, dispose the device's container and keep the USB drive that contains the test data.

Primary objectives:

• Usability evaluation of the FloRite™ system with LUTS patients.

Secondary objectives:

* Comparison of uroflowmetric parameters obtained using home disposable digital uroflowmetry device with standard clinic-based uroflowmetry.
* Evaluation of diurnal variations in uroflowmetric parameters obtained using home uroflowmetry

Primary outcome measures

• Successful use of FloRite™ system in LUTS patients, defined as:

* Successful unpacking and installation
* Successful understanding of the user manual
* Ability of the patients to operate the device as define by a successful test completion and data transmission
* Successful retrieval of the DOK
* Absence of:
* Device dropping down
* Urination outside the container
* Urination on the electronic unit

Secondary outcome measures:

• Comparison of uroflowmetric parameters as measured by

FloRite™ system and standard clinical uroflowmetry as defined by [Time Frame: Days 0, 1, 6 and 7]:

* Qmax - Max Flow Rate

  • Evaluation of diurnal variations in uroflowmetric parameters obtained using home uroflowmetry as defined by [Time Frame: Days 1, 6]:
* Urine flow graph
* Tdelay - Delay time
* T100 - Voiding Time
* TQ - Flow Time
* Tqmax - Time to max Flow
* Qmax - Max Flow Rate
* Qave - Average Flow Rate
* Vcomp - Voided Volume Up to 30 completed patients

Inclusion criteria

* LUTS patients
* Male 18<Age <65
* Ability to speak, read and understand instructions
* Patient willing to sign an Informed Consent Exclusion criteria
* Mentally disabled patients
* Infectious diseases
* Catheterized patients
* Buried penis due to obesity The patients will be consented if found eligible. Prospective, self- controlled, interventional, clinical study

On the baseline visit, after eligibility is confirmed and after consenting the patients, the following steps will be taken:

* Standard clinical uroflowmetry
* Training how to use the system
* Unpacking and setting up the device (supervised by an observer)

The following day, the patient will perform home test with the FloRite™ system. Similar test will be conducted on Day 6 of the study.

The test results will be transferred either by e- mailing the data stored on the DOK or by bringing the DOK itself to the clinic on the 7th day.

On Day 7 of the study, the patients will be asked to return to the clinic for standard clinical uroflowmetry. In addition, the patient will fill a satisfaction questionnaire.

All the measurements must be standard and performed at around the same time.

ELIGIBILITY:
Inclusion Criteria:

* LUTS patients
* Male 18<Age <65
* Ability to speak, read and understand instructions
* Patient willing to sign an Informed Consent

Exclusion criteria:

* Mentally disabled patients
* Infectious diseases
* Catheterized patients
* Buried penis due to obesity

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Usability evaluation of the FloRite™ system with LUTS patients. | Dec-2014
  Primary outcome measures
  • Successful use of FloRite™ system in LUTS patients, defined as:
  * Successful unpacking and installation
  * Successful understanding of the user manual
  * Ability of the patients to operate the device as define by a successful test completion and data transmission
  * Successful retrieval of the DOK
  * Absence of:
  * Device dropping down
  * Urination outside the container
  * Urination on the electronic unit

SECONDARY OUTCOMES:
Comparison of Qmax (Max Flow Rate) | Dec-2014
  Comparison of uroflowmetric parameters of Qmax as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].
Comparison of Tdelay | Dec-2014
  Comparison of uroflowmetric parameters of Tdelay as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].
Comparison of uroflowmetric parameter: T100 - Voiding Time | Dec-2014
  Comparison of uroflowmetric parameters of T100 as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].
Comparison of uroflowmetric parameters of TQ - Flow Time | Dec-2014
  Comparison of uroflowmetric parameters of TQ - Flow Time as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].
Comparison of uroflowmetric parameters of Tqmax - Time to max Flow | Dec-2014
  Comparison of uroflowmetric parameters of Tqmax - Time to max Flow as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].
Comparison of uroflowmetric parameters of Qave | Dec-2014
  Comparison of uroflowmetric parameters of Qave as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].
Comparison of uroflowmetric parameters of Vcomp - Voided volume | Dec-2014
  Comparison of uroflowmetric parameters of Vcomp - Voided volume as measured by FloRite™ system and standard clinical uroflowmetry [Time Frame: Days 0, 1, 6 and 7].

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Leibovitch, Prof., Principal Investigator — Meir Hospital
Locations (1):
- "Meir" Hospital, Kfar Saba, Israel

REFERENCES:
- See also: Sponsor web site. — http://www.flometrica.com